CLINICAL TRIAL: NCT02161419
Title: A Randomized, Double Blind, Placebo-controlled, Multicenter Phase II Study to Evaluate Efficacy and Safety of Roniciclib in Subjects With Extensive-stage Disease Small Cell Lung Cancer (SCLC) Who Are Receiving Cisplatin + Etoposide or Carboplatin + Etoposide as First-line Therapy
Brief Title: RONICICLIB / Placebo in Combination With Chemotherapy in Small Cell Lung Cancer
Acronym: CONCEPT-SCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14615; 2013-004198-28 (EudraCT Number)
Record Dates: First submitted 2014-06-10; First posted 2014-06-11 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Small Cell Lung Carcinoma
Keywords: Small Cell Lung Carcinoma,; First line; Extensive disease; Small cell lung cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — roniciclib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BAY1000394 (Active Comparator): Roniciclib 5 mg bid 3 days on / 4 days off in combination with chemotherapy (carboplatin/etoposide or cisplatin/etoposide) during 6 cycles (21 days each) followed by monotherapy
  Interventions: Drug: Roniciclib (BAY1000394)
- Placebo (Placebo Comparator): Matching placebo 3 days on / 4 days off in combination with chemotherapy (carboplatin/etoposide or cisplatin/etoposide) during 6 cycles (21 days each) followed by monotherapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roniciclib (BAY1000394) — Patients will receive roniciclib treatment as a 3 days on / 4 days schedule off with two 2.5 mg tablets twice daily for a total dose of 10.0 mg/day during 6 cycles (21 days each) of chemotherapy with Carboplatin/etoposide or Cisplatin/etoposide and continue thereafter as monotherapy until tumor progression, unacceptable toxicity, death, consent withdrawal, or withdrawal from the study.
  Arms: BAY1000394
Drug: Placebo — Patients will receive placebo treatment as a 3 days on / 4 days schedule off with two tablets twice daily during 6 cycles (21 days each) of chemotherapy with Carboplatin/etoposide or Cisplatin/etoposide and continue thereafter as monotherapy until tumor progression, unacceptable toxicity, death, consent withdrawal, or withdrawal from the study
  Arms: Placebo

SUMMARY:
This is a study to investigate the potential clinical benefit of roniciclib when given in combination with chemotherapy Carboplatin / Etoposide or Cisplatin / Etoposide as first line treatment in patients with extensive disease small cell lung cancer. Approximately 140 patients will be randomized (1:1) to receive treatment with either roniciclib or placebo in combination with chemotherapy.

Roniciclib is an oral (i.e. taken by mouth) protein kinase inhibitor. A kinase inhibitor targets certain key proteins that are essential for the survival of the cancer cell. The growth of the tumor may be decreased by preventing these specific proteins from functioning. By specifically targeting these proteins, roniciclib in combination with chemotherapy may stop cancer growth.

The primary endpoint (the most meaningful result to be tracked) of this study is based on the progression free survival, i.e. the time the disease is not worsening. The aim is to show that the therapy with roniciclib in combination with chemotherapy prolongs the time the disease is not worsening in this patient population compared to patients receiving placebo in combination with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥18 years (or country-specific legal age of maturity, if >18 years)
* Histologically or cytologically confirmed (extensive-stage disease) ED SCLC (small cell lung cancer)
* At least 1 solid tumor lesion measurable by computer tomography (CT) scan or magnetic resonance imaging (MRI) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1

Exclusion Criteria:

* Prior systemic anticancer therapy for SCLC (including previous therapy with a cyclin-dependent kinase [CDK] inhibitor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2014-07-30 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-05-25 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Up to 17 months

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 17 months
Time to progression (TTP) | Up to 17 months
Overall response rate (ORR) | Up to 17 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (31):
- United States (7):
  - Boca Raton, Florida
  - Port Saint Lucie, Florida
  - St Louis, Missouri
  - Hershey, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Nashville, Tennessee
- Belgium (2):
  - Bruxelles - Brussel
  - Liège
- France (4):
  - Brest
  - Lille
  - Marseille
  - Paris
- Germany (4):
  - Heidelberg, Baden-Wurttemberg
  - Oldenburg, Lower Saxony
  - Essen, North Rhine-Westphalia
  - Großhansdorf
- Hungary (3):
  - Budapest
  - Mátraháza
  - Törökbálint
- Italy (4):
  - Genoa, Liguria
  - Monza-Brianza, Lombardy
  - Sondrio, Lombardy
  - Turin, Piedmont
- Japan (2):
  - Kurume, Fukuoka
  - Bunkyo, Tokyo
- Poland (3):
  - Gdansk
  - Szczecin-Zdunowo
  - Warsaw
- South Korea (2):
  - Seongnam-si, Gyeonggido
  - Seoul

REFERENCES:
- [Derived] Reck M, Horn L, Novello S, Barlesi F, Albert I, Juhasz E, Kowalski D, Robinet G, Cadranel J, Bidoli P, Chung J, Fritsch A, Drews U, Wagner A, Govindan R. Phase II Study of Roniciclib in Combination with Cisplatin/Etoposide or Carboplatin/Etoposide as First-Line Therapy in Patients with Extensive-Disease Small Cell Lung Cancer. J Thorac Oncol. 2019 Apr;14(4):701-711. doi: 10.1016/j.jtho.2019.01.010. Epub 2019 Jan 21. PMID 30677506
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — https://www.clinicaltrialsregister.eu/